CLINICAL TRIAL: NCT07226583
Title: Net-IOB & Exercise Toolkit Pilot Trial: Randomized, Crossover Evaluation of a Behavioral Decision Support Advisor to Improve Glycemic Safety During and After Exercise in Adults With Type 1 Diabetes (NEXT)
Brief Title: Using a Personalized Decision Support Tool to Help People With Type 1 Diabetes Manage Exercise
Acronym: NEXT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: University College Dublin (Other); The Leona M. and Harry B. Helmsley Charitable Trust (Other)
Responsible Party: Principal Investigator, Rayhan A. Lal, Assistant Professor of Medicine & Pediatrics, Stanford University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 82224; 2407-07175 (Other Grant/Funding Number: Leona M & Harry B Helmsley Charitable Trust)
Record Dates: First submitted 2025-10-07; First posted 2025-11-10 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-10

CONDITIONS: Type 1 Diabetes Mellitis; Type 1 Diabetes (T1D); Type 1 Diabetes Mellitus (T1DM)
Keywords: Type 1 Diabetes; T1D; T1DM; Continuous Glucose Monitoring; Insulin Dosing; CGM; Insulin Pump; Exercise; carbohydrate Intake; closed-loop system; hybrid closed-loop
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants complete three supervised exercise visits, each under a different guidance condition (standard-of-care, usual care, or the NEXT decision-support toolkit), in randomized order.
Masking Description: It is not feasible to blind participants or staff to the intervention being applied for each session.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Standard-of-Care (SoC) (Other): Participants follow consensus-based guidance for insulin and carbohydrate adjustments around exercise, as outlined in current international standards. These recommendations are applied by study staff in advance of the exercise session.
  Interventions: Behavioral: Standard-of-Care Guidance (SoC)
- Usual Care (UC) (Other): Participants use their own strategies for managing insulin and carbohydrate around exercise.
  Interventions: Behavioral: Usual Care (UC)
- netIOB & Exercise Toolkit (NEXT) (Experimental): Physicians receive personalized, algorithm-informed recommendations for exercise-related insulin and carbohydrate adjustments. Recommendations are generated using the investigational netIOB & Exercise Toolkit based on CGM data, insulin history, and real-time inputs.
  Interventions: Device: netIOB & Exercise Toolkit (NEXT)

INTERVENTIONS:
Behavioral: Standard-of-Care Guidance (SoC) — Study staff provide insulin and carbohydrate adjustment advice based on consensus exercise management guidelines (Moer et al., 2024), tailored to the planned activity.
  Arms: Standard-of-Care (SoC)
Behavioral: Usual Care (UC) — Participants independently manage their insulin and carbohydrate decisions around exercise, using their routine practices without study-provided guidance.
  Arms: Usual Care (UC)
Device: netIOB & Exercise Toolkit (NEXT) — An investigational software tool generates individualized insulin and carbohydrate adjustment recommendations before and after exercise using CGM data and recent insulin delivery. Study physicians review and relay these recommendations to participants.
  Arms: netIOB & Exercise Toolkit (NEXT)

SUMMARY:
This study evaluates a digital decision-support tool designed to help individuals with type 1 diabetes prepare for exercise. This netIOB & Exercise Tool (NEXT) uses glucose data and insulin delivery history to recommend individualized strategies such as carbohydrate intake, insulin adjustments, or delays in exercise start time.

Participants will complete three structured aerobic or mixed-exercise sessions using different guidance approaches:

(A) published consensus-based standard-of-care guidelines (B) usual personal care routines (C) the NEXT tool

The study compares glucose outcomes, safety, and carbohydrate use across these conditions to inform better exercise preparation and support tools for people with diabetes.

DETAILED DESCRIPTION:
People with type 1 diabetes often experience unpredictable changes in blood glucose levels before, during, and after physical activity. While consensus guidelines exist to help mitigate these risks, many individuals continue to encounter hypoglycemia or rely on excessive carbohydrate intake around exercise.

This study evaluates a software-based tool, netIOB & Exercise Toolkit (NEXT), that provides real-time, individualized guidance for exercise preparation. The tool uses data from continuous glucose monitors (CGMs), insulin delivery history, and exercise timing to suggest adjustments such as carbohydrate intake, temporary targets, or delayed start times. Its goal is to reduce hypoglycemia and carbohydrate burden while preserving exercise safety and feasibility.

The trial uses a randomized, crossover design in which participants complete three supervised moderate-intensity exercise sessions, each under a different preparation strategy. The guidance methods include consensus standard-of-care, usual personal care, and the investigational NEXT tool. Each session is followed for 48 hours to assess glycemic and behavioral outcomes.

Exploratory analyses will stratify glycemic and treatment outcomes based on pre-exercise net insulin-on-board (netIOB) levels, categorized into predefined strata (e.g., 0.0-1.0u, 1.0-2.0u, 2.0-3.0u, 3.0u+), to assess potential effect modification across intervention arms.

The NEXT tool is investigational and classified as IDE-exempt. Findings from this study may inform the design of future clinical trials and support the development of open-source methods for exercise preparation in diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the age of 18-60 years
* Diagnosis of type 1 diabetes for >1 year (based on investigator's clinical judgement)
* Using Tandem Control-IQ and Dexcom G7 for ≥1 month
* Able to sustain moderate intensity walking for 60 minutes (target 50-60% age-predicted HR max) without limitation.
* Use of a stable insulin delivery regimen, with no planned changes in settings or dosing strategy during the study period, and consistent continuous glucose monitor (CGM) use in the prior 1 month (>80% data)

Exclusion Criteria:

* Use of non-continuous subcutaneous insulin infusion (CSII) during study, including long-acting or inhalable insulins.
* Use of other medications with the potential to confound glycemia (including SGLT-2 inhibitors, GIP or GLP-1 receptor agonists) unless on a stable regimen with no planned changes during the study.
* Use of systemic steroids within 4 weeks of planned study participation.
* Severe hypoglycemia (requiring assistance) or DKA within the prior 6 months.
* Intercurrent illness or medical conditions that preclude safe participation in moderate-intensity exercise (e.g. unstable cardiopulmonary disease, uncontrolled arrhythmia, or uncontrolled hypertension), as previously assessed by the individual's primary care physician.
* Pregnancy, lactation, or planned pregnancy during participation.
* Renal insufficiency with eGR <45 mL/min/1.73 m2, dialysis, or adrenal insufficiency.
* Known coronary disease or angina that limits moderate activity, or myocardial infarction/PCI/CABG within 12 months.
* Concurrent participation in another interventional drug/device study within 30 days
* Inability to comply with study procedures or safety requirements (e.g., cannot achieve target HR zone, cannot attend visits, or cannot enable device data access), or otherwise deemed unsuitable by the investigator.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Composite Score of Glycemic Safety and Carbohydrate Burden | Baseline (1 hour pre-exercise), Exercise (0 to 90 minutes), Early Post-Exercise (0 to 6 hours after exercise), Mid Post-Exercise (6 to 24 hours after exercise), Late Post-Exercise (24 to 48 hours after exercise); total of 50.5 hours per visit (3 visits).
  This composite outcome integrates glycemic safety and carbohydrate burden during and after exercise.
  The Glycemic Safety subscore is calculated from percent time spent <70 mg/dl and <54 mg/dl, number of treated hypoglycemic events, and nadir glucose, with heavier penalties for Level 2 hypoglycemia.
  The Carbohydrate Burden Subscore is based on total grams og carbohydrates consumed and the number of treatment episodes.
  A glycemic safety and carbohydrate burden composite metric score of zero is equal to no risk of hypoglycemia without carbohydrate consumption.

SECONDARY OUTCOMES:
Percent-Based Continuous Glucose Monitor Metrics | Baseline (1 hour pre-exercise), Exercise (0 to 90 minutes), Early Post-Exercise (0 to 6 hours after exercise), Mid Post-Exercise (6 to 24 hours after exercise), Late Post-Exercise (24 to 48 hours after exercise); total of 50.5 hours per visit (3 visits).
  Assess standard continuous glucose monitoring (CGM) metrics during defined time windows relative to exercise (0-90 minutes, 0-6 hours, 6-24 hours, and 24-48 hours post-exercise).
  These include:
  * Percent Time in Range (TIR): 70-180 mg/dL
  * Percent Time Below Range (TBR): <70 mg/dL and <54 mg/dL
  * Percent Time Above Range (TAR): >180 mg/dL and >250 mg/dL
Glucose Concentration and Variability Metrics from Continuous Glucose Monitor | Baseline (1 hour pre-exercise), Exercise (0 to 90 minutes), Early Post-Exercise (0 to 6 hours after exercise), Mid Post-Exercise (6 to 24 hours after exercise), Late Post-Exercise (24 to 48 hours after exercise); total of 50.5 hours per visit (3 visits).
  Mean glucose level, glucose standard deviation (SD), and coefficient of variation (CV) will be calculated using CGM data collected over defined time periods relative to exercise. These metrics describe overall glycemic variability and will be used to assess the stability of glucose control following each intervention.
  Units of Measure:
  Mean glucose: mg/dL SD: mg/dL CV: %
Frequency of Hypoglycemic Events | Exercise (0 to 90 minutes), Early Post-Exercise (0 to 6 hours after exercise); total of 7.5 hours per visit (3 visits).
  Number of hypoglycemic episodes per participant at thresholds of <70 mg/dL and <54 mg/dL, stratified by treatment arm. Events will be classified as treated or untreated.
Glucose Nadir Value | Exercise (0 to 90 minutes), Early Post-Exercise (0 to 6 hours after exercise); total of 7.5 hours per visit (3 visits).
  Lowest glucose value (nadir mg/dl) recorded per participant during exercise period and 0-6 hours post-exercise, as measured by CGM.
Time to First Hypoglycemic Event | Exercise (0 to 90 minutes), Early Post-Exercise (0 to 6 hours after exercise); total of 7.5 hours per visit (3 visits).
  Time (in minutes) from exercise start to the first hypoglycemic episode (<70 mg/dL) for each participant.
Carbohydrate Consumption for Hypoglycemia Prevention/Treatment | Exercise (0 to 90 minutes); total of 1.5 hours per visit (3 visits).
  Quantify carbohydrate use related to exercise using:
  * Total grams of carbohydrate consumed
  * Number of carbohydrate treatment episodes
  * Categorization as prophylactic or reactive
Total and Programmed Insulin Delivery | Baseline (1 hour pre-exercise), Exercise (0 to 90 minutes), Early Post-Exercise (0 to 6 hours after exercise), Mid Post-Exercise (6 to 24 hours after exercise), Late Post-Exercise (24 to 48 hours after exercise); total of 50.5 hours per visit (3 visits).
  Compare the total insulin delivered (actual) to the amount that would have been delivered based on the participant's pre-programmed basal rates. This includes both basal and bolus insulin.
Frequency of User-Initiated Pump Adjustments | Baseline (1 hour pre-exercise), Exercise (0 to 90 minutes), Early Post-Exercise (0 to 6 hours after exercise), Mid Post-Exercise (6 to 24 hours after exercise), Late Post-Exercise (24 to 48 hours after exercise); total of 50.5 hours per visit (3 visits).
  Number of times participants manually modified insulin delivery during the exercise period, including suspensions, temporary targets, exercise mode, or basal rate changes.
Duration of User-Initiated Pump Adjustments | Baseline (1 hour pre-exercise), Exercise (0 to 90 minutes), Early Post-Exercise (0 to 6 hours after exercise), Mid Post-Exercise (6 to 24 hours after exercise), Late Post-Exercise (24 to 48 hours after exercise); total of 50.5 hours per visit (3 visits).
  Cumulative duration of user-initiated pump modifications, including time spent in temporary targets, pump suspensions, and exercise modes.

CONTACTS AND LOCATIONS:
Overall Officials: Rayhan Lal, MD, Principal Investigator — Stanford University; Dessi dessi@stanford.edu, PhD, Study Director — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant-level data will be shared, including:
  * Continuous glucose monitoring (CGM) metrics from the Dexcom G7 (e.g., time in range, time below/above range, mean glucose, glucose variability)
  * Carbohydrate treatment data (timing, amount, type)
  * Insulin delivery data (e.g., pump settings, suspensions, automated adjustments)
  * Demographic information (e.g., age range, sex, diabetes duration)
  IPD that will not be shared includes:
  * Direct identifiers (e.g., names, exact dates of birth, addresses)
  * Free-text responses or notes containing potentially identifiable information
  * Any raw data not essential to the reported outcomes or secondary analyses
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available beginning 18 months after article publication and ending 5 years following article publication.
Access Criteria: Proposals should be directed to dessi@stanford.edu. To gain access, data requestors will need to sign a data access agreement.